CLINICAL TRIAL: NCT00710229
Title: A Randomized Observer and Subject Masked Trial Comparing the Visual Outcome After Treatment With Ranibizumab or Bevacizumab in Patients With Neovascular Age-related Macular Degeneration Multicenter Anti VEGF Trial in Austria (MANTA)
Brief Title: Manta Study: Avastin Versus Lucentis in Age Related Macular Degeneration
Acronym: MANTA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Collaborators: Krankenanstalt Rudolfstiftung (Unknown); Medical University of Vienna (Other); Medical University of Graz (Other); Medical University Innsbruck (Other); Krankenhaus der Barmherzigen Brüder Linz (Other); Universitätsaugenklinik Salzburg (Unknown); Hospital Hietzing (Other); Hanuschkrankenhaus (Unknown)
Responsible Party: Susanne Binder Prof, The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK 07-192-1007
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Age Related Macular Degeneration
Keywords: age related macular degeneration; Ranibizumab-Lucentis; Bevacizumab-Avastin
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Intravitreal injectin of Ranibizumab (3 monthly injection followed by monthly injectins as long as required
  Interventions: Drug: Ranibizumab
- B (Active Comparator): Intravitreal injectin of Bevacizumab (3 monthly injection followed by monthly injectins as long as required
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Ranibizumab — intravitreal injection
  Other Names: Lucentis
  Arms: A
Drug: Bevacizumab — intravitreal injection
  Other Names: Avastin
  Arms: B

SUMMARY:
Angiogenesis plays a key role in the development of choroidal neovascularizations (CNV) in age-related macular degeneration. Vascular endothelial growth factor (VEGF) is the most important factor involved in this angiogenetic processes in the eye. This forms the basis for new therapeutic interventions in exudative AMD. Currently two drugs have been approved by the FDA and one drug is used off-label. All these drugs are administered intravitreally. The present study aims to directly compare the effects ranibizumab and bevacizumab in a randomized controlled study in patients with neovascular AMD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Active primary or recurrent subfoveal lesion with CNV secondary to AMD

Exclusion Criteria:

Prior treatment with any intravitreal drug in the study eye

* Prior treatment with verteporfin photodynamic therapy in the study eye
* Prior treatment with systemic bevacizumab
* Prior treatment with any intravitreal durg or verteprofin photodynamic therapy in the nonstudy eye within the 3 moths before the study entry
* Laser photocoagulation within 1 month before study entry in the study eye
* Previous participation in any clinical trial within 1 month before the entry of the study
* Subfoveal fibrosis or atrophy in the study eye
* CNV in either of the two eye due to causes other than AMD such as histoplasmosis or pathologica myopia
* Retinal pigment epithelial tear involving the macula in the study eye
* Any concurrent intraocular condition in the study eye that could either require medical or surgical intervention during the 12 month study period or that could contribute to a loss of best corrected visual acuity over the 12 months study period (e.g. diabetic retinopathy, cataract, uncontrolled glaucoma). The decision on exclusion is to be based on the opinion of the local principal investigator.
* Active intraocular inflammation
* Vitreous hemorrhage in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Change of visual acuity over time | 12 months

SECONDARY OUTCOMES:
Adverse events retinal thickness (OCT) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ludwig Boltzmann Institute for Retinology and Biomicroscopic Lasersurgery, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Krebs I, Schmetterer L, Boltz A, Told R, Vecsei-Marlovits V, Egger S, Schonherr U, Haas A, Ansari-Shahrezaei S, Binder S; MANTA Research Group. A randomised double-masked trial comparing the visual outcome after treatment with ranibizumab or bevacizumab in patients with neovascular age-related macular degeneration. Br J Ophthalmol. 2013 Mar;97(3):266-71. doi: 10.1136/bjophthalmol-2012-302391. Epub 2013 Jan 3. PMID 23292928